CLINICAL TRIAL: NCT05696119
Title: Implementing Injury Prevention Training in Youth Handball (I-PROTECT) Using the RE-AIM Evaluation Framework: A Cluster-randomized Trial
Brief Title: Implementing Injury Prevention Training in Youth Handball (I-PROTECT) Using the RE-AIM Evaluation Framework
Acronym: I-PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-06148-02; 2014/713 (Other: Regional Ethical Review Board in Lund, Sweden)
Record Dates: First submitted 2022-12-13; First posted 2023-01-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Athletic Injuries; Health Behavior
Keywords: Physical activity; Preventive therapy; Adolescent; Health plan implementation; Behaviour change
MeSH Terms: conditions — Athletic Injuries; Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster-randomized study
Who Masked: Outcomes Assessor
Masking Description: An independent statistician, blinded to group allocation, will analyze data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PROTECT (Experimental): I-PROTECT includes physical and psychological injury prevention information and training (i.e., the intervention) and tailored support to implement it specifically developed for Swedish community youth handball.
  Interventions: Behavioral: I-PROTECT
- Control group (Active Comparator): Coaches of youth teams in the control group clubs will be offered currently available injury prevention training (i.e., "Redo för Handboll", English: "Ready for Handball"), accessible online through the Swedish Handball Federation's coach education material.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: I-PROTECT — I-PROTECT is based on existing research and knowledge of experts in sport medicine, sport psychology and implementation science, with the involvement of end-users throughout the process. The interdisciplinary intervention includes end-user-targeted information and injury prevention physical and psychological training, specifically tailored for youth handball. The intervention is delivered through a mobile application (I-PROTECT GO) specifically developed for the I-PROTECT project, including coach, player, club administrator, and caregiver modules. Tailored support to implement I-PROTECT is specifically developed for Swedish community youth handball.
  Arms: I-PROTECT
Behavioral: Control — Coaches of youth teams in the control group clubs will be offered currently available injury prevention training (i.e., "Redo för Handboll", English: "Ready for Handball"), accessible online through the Swedish Handball Federation's coach education material.
  Arms: Control group

SUMMARY:
The aim of this two-armed cluster-randomized controlled trial is to investigate the implementation of the I-PROTECT using the RE-AIM evaluation framework that addresses five dimensions of effectiveness and implementation of interventions: reach, effectiveness, adoption, implementation, and maintenance.

DETAILED DESCRIPTION:
The 'Implementing injury Prevention training ROutines in TEams and Clubs in youth Team handball (I-PROTECT)' project was initiated through dialogue between end-users and researchers with the goal of making injury prevention training an integral part of regular practice in youth handball through a series of studies. Numerous implementation barriers and facilitators were identified in previous studies within the I-PROTECT project. These determinants were addressed when designing the intervention.

The current study was planned with the Swedish Handball Federation, an organization with overall responsibility for handball in Sweden, to investigate whether I-PROTECT will work under real-world conditions and become part of regular handball practice. The specific aim is to investigate the implementation of I-PROTECT using the RE-AIM evaluation framework that addresses five dimensions of effectiveness and implementation of interventions: reach, effectiveness, adoption, implementation, and maintenance. Reach (R) is the absolute number, proportion and representativeness of individuals who are willing to participate in a given intervention. Effectiveness (E) is the impact of the intervention on outcomes. Adoption (A) is the absolute number, proportion and representativeness of settings and intervention agents who are willing to use the intervention. Implementation (I) refers to the intervention agents' fidelity to the various elements of the intervention's protocol. Maintenance (M) is the extent to which the intervention is sustained over time.

The design will be a pragmatic two-armed cluster-randomized controlled trial (cluster-RCT) conforming to the Consolidated Standards of Reporting Trials (CONSORT) statement extension to cluster-randomized trials. Eighteen randomly selected clubs in Sweden offering handball for both female and male youth players, will be randomized to intervention (I-PROTECT) or control (currently available injury prevention training). Implementation outcomes will be investigated using RE-AIM evaluation framework, collected using a study-specific questionnaire at the end of the season (approx. 9 months after study start).

ELIGIBILITY:
Stakeholders (players, coaches, caregivers, club administrators) of all youth teams in randomly selected community handball clubs will be eligible for participation.

Inclusion Criteria:

* Clubs: Clubs in Sweden offering handball for both female and male youth players
* Teams: Training ≥2 times per week
* Youth players: Playing in boys' or girls' teams aged 12-16 years season 2023/2024
* Coaches: leading ≥1 training session/week
* Parents/guardians: directly associated with the eligible players
* Club administrators: engaged in the issues of sports injury, coach education or policy development for youth players

Exclusion Criteria:

* Clubs with previous involvement in developing and/or testing I-PROTECT
* Clubs that offer handball exclusively for either female or male players
* Teams with players 17 years or older

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4225 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Reach as measured by absolute number and proportion of individuals who participate | 9-month follow-up
  Reach outcomes will be: Proportion of eligible stakeholders that register to use the app (players, coaches, club administrators, caregivers), consent to participate (coaches, club administrators), attend online education (coaches, club administrators), and/or respond to a questionnaire (players, coaches, club administrators).
Effectiveness as measured by risk perception | 9-month follow-up
  Risk perception (overall injury risk) is measured on a 7-point rating scale (from extremely low to extremely high) aligned with the Health Action Process Approach (HAPA) (players, coaches, club administrators)
Effectiveness as measured by outcome expectancies | 9-month follow-up
  Outcome expectancies (how preventable injuries are) is measured on a 7-point rating scale (from extremely not preventable to extremely preventable) aligned with the Health Action Process Approach (HAPA) (players, coaches, club administrators)
Effectiveness as measured by perceived effectiveness | 9-month follow-up
  Perceived effectiveness (whether intervention has improved condition/behavior) is measured on a 5-point rating scale (from strongly disagree to strongly agree) from the generic form of the theoretical framework of acceptability (TFA) questionnaire (players, coaches, club administrators)
Adoption as measured by use | 9-month follow-up
  Adoption is measured as having used any components and/or exercises (yes/no) (players, coaches, club administrators)
Adoption as measured by affective attitude | 9-month follow-up
  Affective attitude to intervention is measured on a 5-point rating scale (from strongly dislike to strongly like) from the TFA questionnaire (players, coaches, club administrators)
Adoption as measured by intervention coherence | 9-month follow-up
  Intervention coherence (participant understands how intervention works) is measured on a 5-point rating scale (from strongly disagree to strongly agree) from the TFA questionnaire (coaches, club administrators)
Adoption as measured by self-efficacy | 9-month follow-up
  Self-efficacy (confidence about using intervention) is measured on a 5-point rating scale (from very unconfident to very confident) from the TFA questionnaire (players, coaches, club administrators)
Adoption as measured by burden | 9-month follow-up
  Burden to use intervention is measured on a 5-point rating scale (from no effort at all to huge effort) from the TFA questionnaire (coaches, club administrators)
Adoption as measured by opportunity costs | 9-month follow-up
  Opportunity costs (whether intervention interfered with other priorities) is measured on a 5-point rating scale (from strongly disagree to strongly agree) from the TFA questionnaire (coaches, club administrators)
Adoption as measured by ease of use | 9-month follow-up
  Ease of use is measured on a 5-point rating scale (from strongly disagree to strongly agree) (players, coaches, club administrators)
Implementation as measured by adherence | 9-month follow-up
  Adherence (frequency) of using intervention (players, coaches, club administrators)
Implementation as measured by fidelity to program | 9-month follow-up
  Fidelity to program, i.e. the proportion and type of exercises (players, coaches)
Implementation as measured by fidelity to implementation checklist | 9-month follow-up
  Fidelity to implementation checklist, i.e. proportion of use (club administrators)
Implementation as measured by coping planning | 9-month follow-up
  Plan to deal with challenges is measured on a 7-point rating scale (from extremely disagree to extremely agree) aligned with the Health Action Process Approach (HAPA) (coaches, club administrators)
Maintenance as measured by intention | 9-month follow-up
  Intention to use intervention in the future is measured on a 7-point rating scale (from extremely not likely to extremely likely) aligned with the Health Action Process Approach (HAPA) (players, coaches, club administrators)
Maintenance intention as measured by self-efficacy | 9-month follow-up
  Maintenance self-efficacy (confidence about continuing to use intervention) is measured 7-point rating scale (from extremely not confident to extremely confident) aligned with the Health Action Process Approach (HAPA) (coaches, club administrators)

SECONDARY OUTCOMES:
Implementation determinants | After follow-up, approx. 10 months after study start
  Data will be gathered (e.g., workshops) to enable an in-depth understanding of potential and actual barriers and facilitators, acceptability, usability, and sustainability of I-PROTECT, including its packaging.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ageberg, PhD, Principal Investigator — Lund University
Locations (1):
- Eva Ageberg, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
The current approval by the Regional Ethical Review Board in Lund, Sweden (2014/713, 2020-02952, 2022-06148-02) does not include data sharing. A minimal data set could be shared by request from a qualified academic investigator for the sole purpose of replicating the present study, provided the data transfer is in agreement with EU legislation on the general data protection regulation and approval by the Swedish Ethical Review Authority.
  Contact information:
  Department of Health Sciences, Lund University Box 157, 221 00 Lund, Sweden Contact address: DHSdataaccess@med.lu.se
  Principal Investigator: Eva Ageberg, Department of Health Sciences, Lund University Box 157, 221 00 Lund, Sweden. Email: eva.ageberg@med.lu.se
  Swedish Ethical Review Authority, Box 2110, 75 002 Uppsala, Sweden. Phone: +46 10 475 08 00.

REFERENCES:
- [Derived] Ageberg E, Donaldson A, Strom A, Lucander K, Moesch K, Bunke S, Linnell J, Wedberg R, Ekberg P, Nilsen P. Implementing injury prevention training in youth handball (I-PROTECT) in Sweden: study protocol for a cluster randomised trial. BMJ Public Health. 2024 Jul 30;2(1):e000991. doi: 10.1136/bmjph-2024-000991. eCollection 2024 Jun. PMID 40018138
- See also: Ageberg et al. Implementing injury prevention training in youth handball (I-PROTECT) in Sweden: Study protocol for a cluster-randomized trial — https://bmjpublichealth.bmj.com/content/2/1/e000991